CLINICAL TRIAL: NCT01220193
Title: Evaluation of RTVue in Corneal Measurement
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Qienyuan Zhou, PhD, Optovue
Other Study IDs: RTVue 100 - 2009
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Normal Cornea; Post Laser Refractive Surgery; Cornea Pathology; Cataract Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Normal cornea
- Post laser refractive surgery
- Cornea pathology
- Cataract surgery

SUMMARY:
The purpose of this study is to evaluate RTVue measurement of the cornea in various ocular conditions to include normal, pathology, post refractive surgery and cataract.

ELIGIBILITY:
Inclusion Criteria:

Normal cornea:

* 18 years of age or older
* No corneal pathology
* No prior ocular surgery and no prior laser refractive surgery

Post laser refractive surgery:

* 18 years of age or older
* No corneal pathology
* No prior ocular surgery except laser refractive surgery
* At least 1 week post laser refractive surgery without complication

Corneal pathology:

* 18 years of age or older
* Clinical diagnosis of one or more type of corneal pathologies, including corneal scar and keratoconus, etc., excluding eyes in which corneal power measurement are not clinically relevant (e.g., eyes requiring corneal transplant)
* No prior laser refractive surgery

Cataract surgery:

* 18 years of age or older
* No corneal pathology
* No prior ocular surgery, no prior laser refractive surgery, and no prior cataract surgery
* Post surgery visit shall only include eyes without complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Various ocular conditions to include normal, pathology, post refractive surgery and cataract.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Gordon Binder & Weiss Vision Institute, San Diego, California
  - Brass Eye Center, Latham, New York